CLINICAL TRIAL: NCT01859598
Title: A Prospective, Observational Registry Study Focusing on the Real World Use, Effectiveness and Safety of Initial Basal Insulin Regimen in Type 2 Diabetic Patients Uncontrolled by Oral Antidiabetic Drugs in China
Brief Title: Observational Registry for Basal Insulin Treatment Study (ORBIT)
Status: Completed | Type: Observational
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Chinese Diabetes Society (Other)
Responsible Party: Sponsor
Other Study IDs: ORBIT
Record Dates: First submitted 2012-04-13; First posted 2013-05-22 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
Keywords: diabetes; basal insulin; effectiveness and safety; oral antidiabetic drugs; real world clinical practice
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The scientific use of basal insulin is of great help to individuals and the government. However, there are few studies to investigate the real world use, effect, safety and influence factors of basal insulin in China. This study is to evaluate the use of first basal insulin in China patients with type 2 diabetes with inadequate glycemic control on oral antidiabetic agents (OADs) from the naturalistic clinical practice.

DETAILED DESCRIPTION:
This is a 6-month multicentre, observational, prospective, registry study. About 200 hospitals from different parts of China will take part in this study, and about 20,000 patients with type 2 diabetes mellitus (T2DM) who are inadequately controlled with OADs and willing to accept basal insulin (BI) treatment will be consecutively enrolled during a 12 months period.

The study participants will include at baseline (0 month), 3 month and end point (6 month) to collect the study information. The project will probably last for about 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Type 2 diabetic patients
* Taking OADs before inclusion
* Recently tested HbA1c >=7% at the same site within 3 months
* Being suggested by physician to start basal insulin (BI) treatment
* Willing to start and having been prescribed BI treatment
* Willing to join the registry study and sign the informed consent

Exclusion Criteria:

* Diagnosed with type 1 diabetes
* Received any type of insulin in the last 2 years (except for the intermittent use of insulin of less than 1 month each time)
* With any severe health problem, or any other situation judged by the investigator, that is difficult for the 6 months follow-up
* Current or planned pregnant, lactating women
* Involved in other clinical trial simultaneously or at most 1 month before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meet the following criteria, either from in-patient or out-patient department, will have chance to be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 19894 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Prof., Principal Investigator — The George Institute for Global Health, China
Locations (2):
- China (2):
  - Haidian hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Luo Y, Wu H, Liao X, Zhao T, Cui N, Li A, Sun X, Zhang P, Huang Y, Zhang X, Yin H, Ji L. A Guideline-Based Decision Tree Achieves Better Glucose Control with Less Hypoglycemia at 3 Months in Chinese Diabetic Patients. Diabetes Ther. 2021 Jul;12(7):1887-1899. doi: 10.1007/s13300-021-01075-1. Epub 2021 May 29. PMID 34050897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December of 2011 to June 2013 in secondary and tertiary hospitals all over China, including in-patients and out-patients.
Pre-assignment Details: At the baseline stage:
  Patients registered to assess the eligibility(N=19894); Violate inclusion criteria (N=346); Excluded (N=553);
Groups:
- 6-month Follow-up for Basal Insulin Treatment Study (ORBIT): At the baseline stage:
  Patients registered to assess the eligibility(N=19894); Violate inclusion criteria (N=346); Excluded (N=553);
Period: Visit 2 at 3 Months
Arm/Group | 6-month Follow-up for Basal Insulin Treatment Study (ORBIT)
Started | 18995 (At visit 1, patients remained at baseline, N=18995)
Completed | 17253
Not Completed | 1742
Not completed — Lost to Follow-up | 1742
Period: Visit 3 at 6 Months
Arm/Group | 6-month Follow-up for Basal Insulin Treatment Study (ORBIT)
Started | 17253
Completed | 16341 (Loss to follow-up, N=1517; Come back at visit 3, N=605;)
Not Completed | 912

BASELINE CHARACTERISTICS:
Groups:
- Follow up for 6 Months: At the baseline stage:
  Patients registered to assess the eligibility(N=19894); Violate inclusion criteria (N=346); Excluded (N=553);
Arm/Group | Follow up for 6 Months
Number analyzed (Participants) | 18995
Age, Continuous [Mean (Standard Deviation); unit: year] | 55.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9027
  Male | 9968
Region of Enrollment [Number; unit: participants]
  China | 18995
HbA1c level [Mean (Standard Deviation); unit: %] | 9.6 (2.0)
Fasting Plasma Glucose (FPG) level [Mean (Standard Deviation); unit: mmol/L] | 11.7 (4.0)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.4 (5.3)
Education [Number; unit: participants]
  Primary school or illiterate | 5154
  High school | 10583
  College or higher | 3258
Complication [Number; unit: participants]
  yes | 6744
  no | 12251
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 130.1 (16.0)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 79.5 (9.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.7 (3.4)
Recruitment settings [Number; unit: participants]
  Out-patient | 8361
  In-patient | 10634
Hospital levels [Number; unit: participants]
  Secondary hospitals | 9443
  Tertiary hospitals | 9552
Current residence of patients [Number; unit: participants]
  Urban | 13019
  Rural | 5976
Pre-insulin hypoglycemia [Mean (Standard Deviation); unit: times/person/year] | 1.7 (10.4)
Physical activity [Mean (Standard Deviation); unit: days] | 5.4 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Change in HbA1c During the 6 Months Follow-up.
Description: • Change of HbA1c from baseline to the end-point (6 month).
Time Frame: Baseline and 6 months
Population: the patients who have the results of HbA1c
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Basal Insulin Treatment Study (ORBIT)
Number analyzed (Participants) | 16271
percent | 2.1 (2.1)

2. Primary Outcome: the Change of Hypoglycemia During Follow-up.
Description: •The rate of hypoglycemia at baseline, 3 months (visit 2) and 6 months (visit 3)
Time Frame: baseline and 6 months
Population: The population at visit 3 were used to analyze the hypoglycemia and weight change from visit 1 to visit 3
Measure: Number; unit: percentage of patients with hypoglycemia
Groups:
- Follow up for 6 Months: At the baseline stage:
  Patients registered to assess the eligibility(N=19894); Violate inclusion criteria (N=346); Excluded (N=553);
  At visit 1: Patients remained at baseline, N=18995; Loss to follow-up, N=1742 At visit 2, N=17253; Come back at visit 3, N=605 Loss to follow-up, N=1517 At visit 3, N=16341
Arm/Group | Follow up for 6 Months
Number analyzed (Participants) | 16341
percentage of patients with hypoglycemia
  Visit 1 | 5.6
  visit 2 | 9.6
  visit 3 | 9.0

3. Secondary Outcome: the FPG Change From Visit 1 to Visit 3
Description: the FPG change = the FPG level at visit 1- the FPG level at visit 3
Time Frame: baseline and 6 months
Population: the population in the visit 3 were used for analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Follow up for 6 Months
Number analyzed (Participants) | 16341
mmol/L | 3.8 (4.2)

4. Secondary Outcome: the FPG Control Rate at Visit 3
Description: the percentage of patients who had the FPG level <7.0 mmol/L at visit 3
Time Frame: 6 months
Population: At visit 3, the patients who self-reported their FPG level were used for analysis
Measure: Number; unit: percentage of patients with FPG<7.0
Groups:
- Follow up for 6 Months: At the baseline stage:
  Patients registered to assess the eligibility(N=19894); Violate inclusion criteria (N=346); Excluded (N=553);
  At visit 1: Patients remained at baseline, N=18995; Loss to follow-up, N=1742 At visit 2, N=17253; Come back at visit 3, N=605 Loss to follow-up, N=1517 At visit 3, N=16341, among them, 10416 patients had FPG information
Arm/Group | Follow up for 6 Months
Number analyzed (Participants) | 10416
percentage of patients with FPG<7.0 | 42.5

5. Secondary Outcome: Overall Weight Gain From Visit 1 to Visit 3
Description: the weight gain= the mean weight at visit1 - the mean weight at visit 3
Time Frame: baseline and 6 months
Population: Patients at visit 3 were used for analyzing the change of weight
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Follow up for 6 Months
Number analyzed (Participants) | 16341
Kg | 0.1 (2.94)

ADVERSE EVENTS:
Time Frame: From baseline to 6 months
Description: Led to death; Resulted in a life-threatening illness or injury; Required in-patient hospitalization or prolongation of existing hospitalization; Resulted in permanent impairment of a body structure or function; Led to congenital abnormality or birth defect. Resulted in important medical event or reaction
Arm/Group | Follow up for 6 Months
Serious Adverse Events (participants affected / at risk) | 635/18995
Other Adverse Events (participants affected / at risk) | 0/18995
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follow up for 6 Months (N=18995)
nephroma (Renal and urinary disorders) | 65 (65)
Cardio-cerebrovascular disease (Cardiac disorders) | 258 (258)
pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 103 (103)
nerve system (Nervous system disorders) | 50 (50)
eye disease (Eye disorders) | 23 (23)
Gastrointestinal disease (Gastrointestinal disorders) | 91 (91)
Hepatobiliary disease (Hepatobiliary disorders) | 45 (45)

LIMITATIONS AND CAVEATS:
The characteristics of patients receiving different treatment modalities may not be consistent, and the use of Basal Insulin (BI) depended on individual choices of doctors and patients, resulting in differences in insulin usage among various regions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No